CLINICAL TRIAL: NCT00254124
Title: Efficacy of a Food Portion Control Tool to Induce Weight Loss and Decrease Hypoglycemic Medication Requirements Amongst Obese Type 2 Diabetics.
Brief Title: Use of a Portion Control Food Tool to Induce Weight Loss in Obese Type 2 Diabetics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Stewart Diabetes Education Fund (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17585 (Grant ID#)
Record Dates: First submitted 2005-11-09; First posted 2005-11-15 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: obesity; type 2 diabetes mellitus; portion control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

INTERVENTIONS:
Device: The Diet Plate (R) TM portion control plate and bowl

SUMMARY:
The purpose of this study was to determine whether a food portion control tool would be effective to result in weight loss in a group of overweight type 2 diabetics. We hypothesized that this tool would be effective to induce weight loss in these patients. We also hypothesized that diabetic control would be improved in patients using these plates.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing worldwide. Portion size is known to be an important determinant of energy intake. However, to our knowledge, no clinical trials have previously been conducted which examine the efficacy of a food portion control tool to control caloric intake and thereby induce weight loss.

Most cases of type 2 diabetes can be attributed directly to obesity. Dietary caloric restriction has been shown to improve glycemic control by virtue of weight loss, with an additional benefit independent of weight loss.

Comparison: daily use of a food portion control tool plus usual care at a diabetes care center, compared to usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosis of type 2 diabetes mellitus
* body mass index of 30 or greater
* a member of the Diabetes Education Center in Calgary, AB, Canada, for at least 6 months prior to study enrollment

Exclusion Criteria:

* taking a weight loss medication (sibutramine or orlistat)
* weight loss >10 lbs in 2 months preceding study enrolment
* consumption of dinner at restaurants more than twice weekly
* current diagnosis of cancer
* psychiatric illness under care of a psychiatrist
* surgery in the 3 months prior to the study, or expected during the study period
* history of bulimia or anorexia nervosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2004-04; Study Completion 2004-12

PRIMARY OUTCOMES:
- percentage change in body weight
- proportion of each group that achieve a clinically significant (>=5%) reduction in body weight
- prespecified per protocol analysis: same outcomes as above, looking at patients who were >=80% compliant with the intervention

SECONDARY OUTCOMES:
- change in glycosylated hemoglobin
- change in serum cholesterol
- change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Sue D Pedersen, MD, FRCPC, Study Director — Division of Endocrinology and Metabolism, University of Calgary, Calgary, AB, Canada; Greg A Kline, MD, FRCPC, Principal Investigator — Division of Endocrinology and Metabolism, University of Calgary, Calgary, AB, Canada
Locations (1):
- Diabetes Education Center, Colonel Belcher Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Pedersen SD, Kang J, Kline GA. Portion control plate for weight loss in obese patients with type 2 diabetes mellitus: a controlled clinical trial. Arch Intern Med. 2007 Jun 25;167(12):1277-83. doi: 10.1001/archinte.167.12.1277. PMID 17592101